CLINICAL TRIAL: NCT00775554
Title: "Are Ultrasound-guided Hematoma Blocks for Distal Forearm Fractures Superior to the Landmark-guided Method for Hematoma Blocks?"
Brief Title: Comparison Study of Using Ultrasound Guidance for Hematoma Blocks vs. Traditional Approach
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-118
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2008-10

CONDITIONS: Forearm Fracture
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional hematoma block (Other): people will receive traditional hematoma block for closed forearm fractures
  Interventions: Other: ultrasound guided hematoma block
- ultrasound guided hematoma block (Other): pts. will receive a hematoma block using bedside ultrasound to guide the placement
  Interventions: Other: ultrasound guided hematoma block

INTERVENTIONS:
Other: ultrasound guided hematoma block — pt. will receive ultrasound guided hematoma block
  Other Names: ultrasound
  Arms: traditional hematoma block
Other: ultrasound guided hematoma block — ultrasound will be used to guide hematoma blocks
  Other Names: ultrasound
  Arms: ultrasound guided hematoma block

SUMMARY:
Will use visual analog scales to compare effectiveness of traditional hematoma block vs ultrasound guided hematoma block with regards to pain. This will be done for closed forearm fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Closed forearm fracture

Exclusion Criteria:

* Mentally impaired, visually impaired or deaf
* Age < 18
* Alcohol on board

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale movement

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Roosevelt Hospital, New York, New York, United States